CLINICAL TRIAL: NCT01943994
Title: Psilocybin-facilitated Smoking Cessation Treatment: A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Beckley Foundation (Other); Heffter Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NA_00016166
Record Dates: First submitted 2013-09-12; First posted 2013-09-17 (Estimated); Results first posted 2024-07-24 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Nicotine Dependence
Keywords: Psilocybin; Smoking cessation
MeSH Terms: conditions — Tobacco Use Disorder; Smoking Cessation | interventions — Nicotine Replacement Therapy; Tobacco Use Cessation Devices; Nicotine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Psilocybin-assisted treatment (Experimental): Participants will receive a 13-week cognitive behavioral intervention for smoking cessation, with a high dose of psilocybin (30mg / 70kg) to be administered on the Target Quit Date in week 5.
  Interventions: Drug: Psilocybin-assisted treatment
- Nicotine Replacement Therapy (NRT) (Active Comparator): Participants will receive a 13-week cognitive behavioral intervention for smoking cessation, with a standard 8 to 10-week regimen of NRT to be administered beginning on the Target Quit Date in week 5. NRT for this study will be a transdermal nicotine patch administered according to recommended label usage (For individuals who smoke more than 10 cigarettes per day: 21mg daily weeks 1-6, 14mg daily weeks 7-8, 7mg daily weeks 9-10. For individuals who smoke 10 or less cigarettes per day: 14mg daily for weeks 1-6, 7mg daily for weeks 7-8).
  Interventions: Drug: Nicotine Replacement Therapy (NRT)

INTERVENTIONS:
Drug: Psilocybin-assisted treatment — Participants will be administered 30 mg/70 kg psilocybin. Preliminary evidence from our ongoing psilocybin dose-effects study suggests that this dose is associated with mystical-type experiences.
  Other Names: O-phosphoryl-4-hydroxy-N,N-dimethyltryptamine
  Arms: Psilocybin-assisted treatment
Drug: Nicotine Replacement Therapy (NRT)
  Other Names: Transdermal Nicotine Patch; Nicoderm CQ
  Arms: Nicotine Replacement Therapy (NRT)

SUMMARY:
One of the most promising lines of investigation for the therapeutic use of hallucinogens in the 1960s and 1970s was in the treatment of drug dependence. The investigators propose to examine psilocybin administration combined with a structured smoking cessation treatment program in nicotine dependent individuals in order to provide preliminary data on the efficacy of this combined treatment for smoking cessation. Prior work in the investigators laboratory has shown that under carefully prepared and supportive conditions, psilocybin administration can facilitate highly salient experiences with enduring personal meaning and spiritual significance. It is plausible that embedding such highly meaningful experiences into a drug dependence cessation attempt may provide an enduring motivation for remaining abstinent. Cigarette smoking is a good model system for studying drug dependence because users are less likely to be challenged by the many social and economic impairments that often accompany dependence on other drugs such as cocaine, heroin, or alcohol. More specifically, the investigators propose to conduct a randomized controlled comparative efficacy study in which either psilocybin or transdermal nicotine patch are administered under highly supportive conditions to individuals who are nicotine-dependent cigarette smokers, who have had multiple unsuccessful quit attempts, and who continue to desire to quit smoking. Other than nicotine dependence, participants will be healthy. Fifteen participants have already completed a preliminary open-label pilot-study with no control condition. Eighty additional participants will be enrolled and randomized to either psilocybin (n=40), or nicotine patch (n=40) treatment. Participants will receive a 13-week course of cognitive behavioral therapy for smoking cessation, with Target Quit Date set for week 5. After several preparation meetings with study monitors, participants will have either a single day-long psilocybin session using a high dose (30 mg/70 kg), or a standard 8 to 10-week course of nicotine patch treatment. Participant smoking status will be assessed repeatedly for 8 weeks after the Target Quit Date, including biological verification of smoking status through breath and urine samples. Smoking status will also be assessed at three follow up sessions approximately 3, 6, and 12 months after the Target Quit Date. Additionally, 50 of these participants (25 per treatment condition) will undergo MRI scanning before and after Target Quit Date to assess the brain-based mechanisms associated with these treatments. Individuals assigned to the nicotine patch study treatment condition will be eligible to undergo an optional high dose psilocybin session after completing the 6-month follow-up meeting.

ELIGIBILITY:
Inclusion Criteria:

* 21 to 65 years old.
* Have given written informed consent.
* Have a high school level of education.
* Be a daily smoker with multiple unsuccessful previous quit attempts, and report a continued desire to quit smoking.
* Agree to abstain from smoking and alcohol for 24-hours, and caffeine for 12-hours prior to MRI scanning (for MRI participants only).
* Agree to abstain from smoking for the psilocybin session from 1 hour before psilocybin administration until at least 30 hours afterwards.
* Agree to consume approximately the same amount of caffeine-containing beverage (e.g., coffee, tea) that he/she consumes on a usual morning, before arriving at the research unit on the morning of drug session day. If the volunteer does not routinely consume caffeinated beverages, he or she must agree not to do so on session day.
* Agree to refrain from using any psychoactive drugs, including alcoholic beverages, within 24 hours of psilocybin administration. Exceptions include caffeine and nicotine.
* Be healthy as determined by screening for medical problems via a personal interview, a medical questionnaire, a physical examination, an electrocardiogram (ECG), and routine medical blood and urinalysis laboratory tests.

Exclusion Criteria:

* Women who are pregnant (positive pregnancy test) or nursing, or are not practicing an effective means of birth control
* Cardiovascular conditions: uncontrolled hypertension, angina, a clinically significant ECG abnormality (e.g., atrial fibrilation), TIA in the last 6 months stroke, peripheral or pulmonary vascular disease
* Epilepsy with history of seizures
* Insulin-dependent diabetes; if taking oral hypoglycemic agent, then no history of hypoglycemia
* Currently taking psychoactive prescription medication on a regular basis
* Currently taking on a regular (e.g., daily) basis any medications having a primary centrally-acting pharmacological effect on serotonin neurons or medications that are MAO inhibitors. For individuals who have intermittent or PRN use of such medications, psilocybin sessions will not be conducted until at least 5 half-lives of the agent have elapsed after the last dose.
* Have HIV or Syphilis.
* Have any current neurological illnesses including, but not limited to, seizure disorders, frequent migraines or on prophylaxis, multiple sclerosis, movement disorders, history of significant head trauma, or CNS tumor.
* Morbidly obese, or severely underweight as determined by medical examination.
* Not suitable to undergo an MRI session due to certain implanted devices (cardiac pacemaker or neurostimulator, some artificial joints, metal pins, surgical clips or other implanted metal parts), body morphology, or claustrophobia (for MRI participants only).
* Current or past history of meeting DSM-IV criteria for Schizophrenia, Psychotic Disorder (unless substance-induced or due to a medical condition), or Bipolar I or II Disorder.
* Current or past history within the last 5 years of meeting DSM-IV criteria for alcohol or drug dependence (excluding caffeine and nicotine) or severe major depression.
* Have a first or second degree relative with schizophrenia, psychotic disorder (unless substance induced or due to a medical condition), or bipolar I or II disorder.
* Currently meets DSM-IV criteria for Dissociative Disorder, Anorexia Nervosa, Bulimia Nervosa, Major Depression, or Post-traumatic Stress Disorder.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2008-09 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-11-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew W Johnson, PhD, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - Behavioral Pharmacology Research Unit, Baltimore, Maryland
  - Neuroimaging Research Branch, NIDA-IRP, Baltimore, Maryland

REFERENCES:
- See also: study recruitment website — https://www.QuitSmokingBaltimore.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Nicotine Replacement Therapy (NRT) First, Then Psilocybin-assisted Treatment: Participants will receive a 13-week cognitive behavioral intervention for smoking cessation, with a standard 8 to 10-week regimen of NRT to be administered beginning on the Target Quit Date in week 5. NRT for this study will be a transdermal nicotine patch administered according to recommended label usage (For individuals who smoke more than 10 cigarettes per day: 21mg daily weeks 1-6, 14mg daily weeks 7-8, 7mg daily weeks 9-10. For individuals who smoke 10 or less cigarettes per day: 14mg daily for weeks 1-6, 7mg daily for weeks 7-8).
  Participants who were initially assigned to the "Nicotine Replacement Therapy (NRT)" Arm/Group had the option to cross-over to "Psilocybin-assisted Treatment" at 6 months.
Period: Period 1: Initial Treatment (6 Months)
Arm/Group | Psilocybin-assisted Treatment | Nicotine Replacement Therapy (NRT) First, Then Psilocybin-assisted Treatment
Started | 42 | 40
Completed | 35 | 34
Not Completed | 7 | 6
Period: Period 2: Optional Cross-over (6 Months)
Arm/Group | Psilocybin-assisted Treatment | Nicotine Replacement Therapy (NRT) First, Then Psilocybin-assisted Treatment
Started | 35 | 34
Participants Who Completed the Optional Cross-over Psilocybin Session | 0 | 26
Completed | 34 | 28
Not Completed | 1 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Psilocybin-assisted Treatment | Nicotine Replacement Therapy (NRT) First, Then Psilocybin-assisted Treatment | Total
Number analyzed (Participants) | 42 | 40 | 82
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 38 | 40 | 78
  >=65 years | 4 | 0 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.48 (11.93) | 46.75 (12.26) | 47.63 (12.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 14 | 33
  Male | 23 | 26 | 49
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 0 | 3
  White | 38 | 35 | 73
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 42 | 40 | 82

OUTCOME MEASURES:

1. Primary Outcome: Prolonged Abstinence: Biologically Verified Cigarette Smoking Abstinence for 6 Months
Description: Cigarette smoking abstinence from the target quit (allowing for an initial 14-day grace period) to the 6-month follow up, as verified by breath carbon monoxide, urine cotinine, and retrospective self-report.
Time Frame: From the target quit date to the 6-month follow up
Measure: Count of Participants; unit: Participants
Groups:
- Nicotine Replacement Therapy (NRT): Participants will receive a 13-week cognitive behavioral intervention for smoking cessation, with a standard 8 to 10-week regimen of NRT to be administered beginning on the Target Quit Date in week 5. NRT for this study will be a transdermal nicotine patch administered according to recommended label usage (For individuals who smoke more than 10 cigarettes per day: 21mg daily weeks 1-6, 14mg daily weeks 7-8, 7mg daily weeks 9-10. For individuals who smoke 10 or less cigarettes per day: 14mg daily for weeks 1-6, 7mg daily for weeks 7-8).
  Nicotine Replacement Therapy (NRT)
Arm/Group | Psilocybin-assisted Treatment | Nicotine Replacement Therapy (NRT)
Number analyzed (Participants) | 42 | 40
Participants | 17 | 4
Statistical Analysis 1: Comparison: Psilocybin-assisted Treatment vs Nicotine Replacement Therapy (NRT); Test type: Superiority; p = 0.003, Regression, Logistic; Odds Ratio (OR) = 6.12, 95% CI 2-sided [1.99 to 23.26]

2. Secondary Outcome: Prolonged Abstinence: Biologically Verified Cigarette Smoking Abstinence for 3 Months
Description: Cigarette smoking abstinence from the target quit (allowing for an initial 14-day grace period) to the 3-month follow up, as verified by breath carbon monoxide, urine cotinine, and retrospective self-report.
Time Frame: From the target quit date to the 3-month follow up
Measure: Count of Participants; unit: Participants
Arm/Group | Psilocybin-assisted Treatment | Nicotine Replacement Therapy (NRT) First, Then Psilocybin-assisted Treatment
Number analyzed (Participants) | 42 | 40
Participants | 20 | 12

3. Secondary Outcome: Prolonged Abstinence: Biologically Verified Cigarette Smoking Abstinence for 12 Months
Description: Cigarette smoking abstinence from the target quit (allowing for an initial 14-day grace period) to the 12-month follow up, as verified by breath carbon monoxide, urine cotinine, and retrospective self-report.
Time Frame: From the target quit date to the 12-month follow up
Population: Participants with data collected
Measure: Count of Participants; unit: Participants
Groups:
- Cross-over to Psilocybin-assisted Treatment: Participants in the Nicotine Replacement Therapy (NRT) arm were also eligible to receive a single high-dose (30mg/70kg) psilocybin administration after completing the primary study endpoint at 6-month follow-up. Thus, individuals in this category opted to complete this cross-over psilocybin session after completing a course of NRT.
Arm/Group | Psilocybin-assisted Treatment | Nicotine Replacement Therapy (NRT) | Cross-over to Psilocybin-assisted Treatment
Number analyzed (Participants) | 42 | 14 | 26
Participants | 15 | 0 | 7

ADVERSE EVENTS:
Time Frame: Up to 12 months
Description: After TQD participants were asked at each study visit about any adverse events (AEs) since their last visit, which were documented, including duration, severity, and relatedness. Participants in the Nicotine Replacement Therapy (NRT) arm were eligible to receive a 30mg/70kg psilocybin session after completing the primary 6-month follow-up. Those who completed this cross-over psilocybin session received 2 interventions (NRT and psilocybin), so their AEs are reported separately.
Arm/Group | Psilocybin-assisted Treatment | Nicotine Replacement Therapy (NRT) | Cross-over to Psilocybin-assisted Treatment
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/40 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/42 | 1/40 | 1/26
Other Adverse Events (participants affected / at risk) | 37/42 | 31/40 | 25/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Psilocybin-assisted Treatment (N=42) | Nicotine Replacement Therapy (NRT) (N=40) | Cross-over to Psilocybin-assisted Treatment (N=26)
Gallstones / gallbladder removal (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Suicidal Ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Psilocybin-assisted Treatment (N=42) | Nicotine Replacement Therapy (NRT) (N=40) | Cross-over to Psilocybin-assisted Treatment (N=26)
Depression (Psychiatric disorders) | 12 (22) | 10 (13) | 2 (3)
Headache (Nervous system disorders) | 22 (24) | 4 (4) | 15 (16)
Elevated Blood Pressure (Cardiac disorders) | 24 (24) | 0 (0) | 15 (15)
Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 9 (12) | 9 (14) | 4 (5)
Anxiety (Psychiatric disorders) | 9 (10) | 12 (13) | 4 (4)
Insomnia (Psychiatric disorders) | 3 (5) | 8 (10) | 3 (3)
GI Illness / Diarrhea (Gastrointestinal disorders) | 9 (10) | 4 (4) | 2 (3)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 7 (9) | 0 (0)
Irritability (Psychiatric disorders) | 4 (6) | 2 (3) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 3 (3) | 2 (2)
Nausea (Gastrointestinal disorders) | 3 (3) | 3 (4) | 3 (4)
Visual Disturbance (Eye disorders) | 5 (7) | 0 (0) | 3 (3)
Vivid Dreams (Psychiatric disorders) | 0 (0) | 6 (7) | 0 (0)
Fatigue (General disorders) | 3 (3) | 2 (3) | 3 (3)
Joint Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4) | 2 (2)
Migraine (Nervous system disorders) | 2 (2) | 1 (3) | 1 (2)
Elevated Heart Rate (Cardiac disorders) | 2 (2) | 2 (3) | 2 (2)
Concentration Impairment (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0)
Fever (General disorders) | 0 (0) | 2 (2) | 0 (0)
Ear Infection (Ear and labyrinth disorders) | 0 (0) | 2 (2) | 0 (0)
Panic (Psychiatric disorders) | 1 (1) | 0 (0) | 3 (3)
Hernia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Emotional Lability (Psychiatric disorders) | 0 (0) | 0 (0) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-04-15): https://cdn.clinicaltrials.gov/large-docs/94/NCT01943994/Prot_SAP_000.pdf